CLINICAL TRIAL: NCT02316405
Title: Can Arm and Leg Cycling Exercise Improve Walking After Stroke?
Brief Title: Can Arm and Leg Cycling Exercise Improve Walking After Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Victoria (Other)
Responsible Party: Principal Investigator, Dr. E. Paul Zehr, Dr. E. Paul Zehr, University of Victoria
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: D015017-2011-2014; 123456 (Other: Heart and Stroke Foundation of Canada)
Record Dates: First submitted 2014-12-09; First posted 2014-12-12 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-12

CONDITIONS: Cerebrovascular Accident
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Test Group (Experimental): 5 weeks of arm and leg cycling, 3 times per week for 30 minute of total exercise per session
  Interventions: Other: Arm and Leg Cycling Exercise for Walking after Stroke

INTERVENTIONS:
Other: Arm and Leg Cycling Exercise for Walking after Stroke

SUMMARY:
It has been found that arm and leg cycling is similar to walking. Thus, the objective of this research is to determine if arm and leg cycling can be used to improve walking ability in a post-stroke population. This outcome would directly impact the health and quality of life for those who have suffered a stroke.

DETAILED DESCRIPTION:
It has been found that arm and leg cycling is similar to walking in terms of the muscle activation patterns, joint ranges of motion, and neural pathways activated. Another advantage of arm and leg cycling is that it involves coordination of all four limbs in a rhythmic movement. This may be particularly beneficial given previous findings that arm movement contributes to the activation of leg muscles during walking in humans. This is achieved with interconnected neural pathways that link the arms to the legs. These neural interlimb connections remain intact in stroke victims, such that maximizing the contribution of the arms to the legs may increase coordination for walking.

Thus, the objective of this research is to determine if arm and leg cycling can be used to increase the strength of inter-limb connections and if this helps to improve walking ability in a post-stroke population. 15-20 participants will be recruited to participate in a five week training intervention where measures will be taken before and after the intervention to assess efficacy. Arm and leg cycling could provide a novel method to improve inter-limb coupling and walking ability. These outcomes would directly impact the health and quality of life for those who have suffered a stroke.

ELIGIBILITY:
Inclusion Criteria:

* Cerebrovascular accident

Exclusion Criteria:

* Inability to stand

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-07; Primary Completion 2014-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Walking Ability | Within five days
  Treadmill test of walking coordination, speed, and symmetry. Interlimb coordination assessed with peripheral nerve stimulation during arm and leg cycling and walking. Strength of dorsi-flexion and plantar-flexion and grip strength also assessed.

SECONDARY OUTCOMES:
Clinical Status assessed by a Physiotherapist | Within 5 days
  Clinical assessment of skin sensitivity, spasticity, balance and coordination, and walking endurance.

CONTACTS AND LOCATIONS:
Overall Officials: E P Zehr, Doctorate, Principal Investigator — University of Victoria
Locations (1):
- MacLaurin Building, Victoria, British Columbia, Canada